CLINICAL TRIAL: NCT06644157
Title: Treatment and Prevention of Melasma Relapses by Using 1064nm 650 Microsecond Laser: a Prospective Randomized Intra-individual Study
Brief Title: Treatment and Prevention of Melasma Relapses by Using 1064nm 650 Microsecond Laser
Acronym: Melasma650
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-PP-02
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Using the Aerolase laser (Experimental): All patients applied to the entire face the cosmetic depigmenting agent Mela B3 (La Roche Posay) cream twice daily for 3 months. One session of laser on one side of the face (randomly assigned for each patient for the duration of the study) will be performed every other week for 12 weeks for a total of 6 sessions. All the patients will apply the entire face a sunscreen of sun protection factor 50 with high UVA protection (UV Mune 400; La Roche Posay) during the entire study duration.
  Interventions: Device: Laser Néo Élite

INTERVENTIONS:
Device: Laser Néo Élite — One session of laser on one side of the face (randomly assigned for each patient for the duration of the study) will be performed every other week for 12 weeks for a total of 6 sessions. All the patients will apply the entire face a sunscreen of sun protection factor 50 with high UVA protection (UV Mune 400; La Roche Posay) during the entire study duration.

SUMMARY:
Melasma is a frequently acquired hyperpigmentary disorder affecting up to 30% of child-bearing women in some populations. Melasma is still often called chloasma or the pregnancy mask and is considered as the main consequence of female hormone stimulation on a predisposed genetic background but only 20% of pregnant women are affected. The investigator hypothesize that the Aerolase laser treatment could not only enhance the efficacy of the topical depigmenting agents but also by reducing the vascular component decrease the intensity of the relapses.

All patients applied to the entire face the cosmetic depigmenting agent Mela B3 (La Roche Posay) cream twice daily for 3 months. One session of laser on one side of the face (randomly assigned for each patient for the duration of the study) will be performed every other week for 12 weeks for a total of 6 sessions. All the patients will apply the entire face a sunscreen of sun protection factor 50 with high UVA protection (UV Mune 400; La Roche Posay) during the entire study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with a clinically diagnosed moderate to severe melasma (mMASI above 5)
2. ≥ 18 years old
3. For Women of childbearing potential (WOCBP), an effective contraception (estroprogestative pill, contraceptive implant, IUD, condoms or tubal ligation) should be used for more than one month before the inclusion in the study.

   Women of childbearing potential (WOCBP) must have a negative urine pregnancy test result at baseline.

   WOCBP are defined as women who are biologically capable of becoming pregnant, including women who are using contraceptives or whose sexual partners are either sterile or using contraceptives.

   Women of non-childbearing potential (WONCBP) do not require a urine pregnancy test and must meet at least one of the following criteria:
   * Have undergone hysterectomy or bilateral oophorectomy.
   * Have medically confirmed ovarian failure; or
   * Are medically confirmed to be post-menopausal (cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause).
4. Affiliation to a social security system
5. Signed informed consent
6. Patient willing and able to attend all study visits

Exclusion Criteria:

1. Pregnant or breast-feeding women or women with potential childbearing and not taking contraceptives or who plan to get pregnant during the study duration.
2. Patient with additional facial pigmentary disorder.
3. Patient having used a depigmenting cosmetic in the month prior to inclusion or having used a local corticosteroid on the skin, eyes, nose or mouth (inhaled corticosteroid) or systemic corticosteroids in the month prior to inclusion or having used local tretinoin or local hydroquinone in the month prior to inclusion.
4. Patient having other facial dermatosis that may interfere with the evaluation of the treatment
5. Patient having used a local corticosteroid on the skin, eyes, nose or mouth (inhaled corticosteroid) or systemic corticosteroids during the month preceding inclusion.
6. Patients with a contraindication to laser treatment are :

   * A history of keloids or other abnormal scars.
   * Use of photosensitising medication or history of photosensitivity disorders - Lupus erythematosus
   * Sunburn in the treatment area
   * Active infection in the treatment area
7. Patient having used local tretinoin or local hydroquinone during the month preceding inclusion.
8. Patient undergoing chronic anti-inflammatory treatment (NSAID use accepted if less than 10 days cumulative over the entire study).
9. Patient with a history of clinically significant allergy, in particular to components of the products studied.
10. Adult under guardianship or deprived of freedom
11. Patient in a situation, which, in the opinion of the Investigator, may interfere with optimal participation in the study.
12. Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation.
13. Patient unable to communicate effectively with Investigator or unable to follow study requirements
14. Patient refusing to be photographed within the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Melasma Area and Severity Index | at 24 weeks
  Evaluation of hemi modified hemi mMASI at week 24 for each laser-treated and not laser-treated areas separately. The score was 0-24.

SECONDARY OUTCOMES:
Satisfaction patient | at week 12
  The patient global assessment is a score graded from 0 (clear); 1 (marked improvement); 2 (moderate improvement); 3 (slight improvement); 4 (no improvement); 5 (worse)

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Passeron, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided